CLINICAL TRIAL: NCT04307589
Title: Healthy Grandparenting: The Impact of Non-residential Grandchild Care on Physical Activity and Sedentary Behavior in People Aged 50 Years and Over
Brief Title: The Impact of Grandchild Care on Physical Activity and Sedentary Behavior in People Aged 50 Years and Over
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Research Foundation Flanders (Other); University Ghent (Other)
Responsible Party: Principal Investigator, Marie Vermote, Principal Investigator, Vrije Universiteit Brussel
Other Study IDs: 2020-067
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Adults Aged 50 Years and Older
Keywords: grandparents; grandchildren; caregiving; physical activity; sedentary behavior; body composition; quality of life; prospective cohort study
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Caregiving grandparents
  Interventions: Other: Observation
- Non-caregiving grandparents
  Interventions: Other: Observation
- Middle-aged and older adults not being a grandparent
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — An observational follow-up study will be implemented over a period of 2 years, consisting of 3 test occasions with a fixed time interval of 1 year in between (T0 = baseline, T1 = 12 months, T2 = 24 months). Data will be collected in participants who provide grandchild care in a non-residential grandparent context as well as in a sample of non-caregiving grandparents and a sample of middle-aged and older adults not being a grandparent. All three samples will thus be prospectively monitored over a period of 2 years.

SUMMARY:
Given the widespread provision of grandparental child care, examining its impact on grandparents' energy-expenditure related behaviors in the broader context of health is imperative. The maintenance of functional independence and good quality of life is critical at a more advanced age. It has been put forward that an increased duration, frequency and intensity of physical activity (PA) combined with a restriction of sedentary behavior (SB) is the most important strategy to reduce morbidity risk and to foster health in an aging population. The present study aims to fill a gap in current knowledge on (changes in) caregiving grandparents' PA levels and SB patterns. An observational follow-up study will be conducted to examine and compare both energy-expenditure related behaviors linked to body composition and health-related quality of life among caregiving grandparents, non-caregiving grandparents and non-grandparent peers, both momentarily and over time. This fundamental research aims to provide scientific evidence contributing to the promotion of healthy grandparenting in people on the threshold of old age in modern society.

DETAILED DESCRIPTION:
The first objective of the study is to provide a detailed overview of habitual levels of physical activity and sedentary behavior among caregiving grandparents in relation to their body composition and health-related quality of life (including both physical and mental function), and to identify to what extent these outcome measures are associated with the number, sex and age of the grandchild(ren) as well as with the intensity of grandparents' provision of child care, while taking some demographic characteristics of the grandparent (i.e., age, sex, marital status, socio-economic status (SES)) into account.

The second objective is to compare caregiving grandparents' energy-expenditure related behaviors (i.e., physical activity and sedentary behavior) and their link with health-related measures of interest (i.e., body composition and quality of life) with both non-caregiving grandparents and non-grandparent peers as relevant control groups.

The third objective is to investigate (age-related) changes in physical activity and sedentary behavior linked to body composition and health-related quality of life among caregiving grandparents versus non-caregiving grandparents as well as non-grandparents both in the short and the longer term, and to identify possible predictors of these changes over time. Additionally, it is the intention to examine the impact of middle-aged and older adults making the transition to (caregiving) grandparenthood on both energy-expenditure related behaviors as well as the health-related measures of interest.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥50 years of age
* Speaking the Dutch language
* Being able to perform independent locomotion (e.g. not relying on a walking aid or wheelchair, etc.)
* Not suffering from a known cognitive impairment affecting one's memory, attention or understanding (e.g. dementia, brain injury, etc.)
* Not living in a residential care center for elderly people

Exclusion Criteria:

* Being <50 years of age
* Not speaking the Dutch language
* Not being able to perform independent locomotion (e.g. relying on a walking aid or wheelchair, etc.)
* Suffering from a known cognitive impairment affecting one's memory, attention or understanding (e.g. dementia, brain injury, etc.)
* Living in a residential care center for elderly people

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People aged 50 years and over with and without grandchildren.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | At baseline (T0), at 12 months (T1), at 24 months (T2)
  Physical activity will be assessed subjectively by using a self-reported questionnaire (International Physical Activity Questionnaire (IPAQ - Dutch version)) and objectively by using a tri-axial accelerometers (Actigraph, wGT3X-BT) over a one-week period.
Change in sedentary behavior | At baseline (T0), at 12 months (T1), at 24 months (T2)
  Sedentary behavior will be assessed subjectively by using a self-reported questionnaire (Sedentary Behavior Questionnaire for (older) adults in Dutch) and objectively by using a tri-axial accelerometers (Actigraph, wGT3X-BT) over a one-week period.

SECONDARY OUTCOMES:
Change in body dimensions | At baseline (T0), at 12 months (T1), at 2 year months (T2)
  Body height measured by means of mobile equipment (SECA 213). Body weight measured by means of mobile equipment (TANITA MC-780 SM A). Waist and hip circumferences will be measured by means of Cescorf measuring tape.
Change in body composition | At baseline (T0), at 12 months (T1), at 2 year months (T2)
  Body composition will be measured by bio-electrical impedance analysis (BIA, TANITA MC-780 S MA) to estimate fat mass, fat free mass and muscle mass.
Change in quality of life: self-reported questionnaire | At baseline (T0), at 12 months (T1), at 24 months (T2)
  Quality of life will be measured subjectively by using a self-reported questionnaire (Multipurpose 36-item Short-Form Health Survey version 2.0 (SF-36v2) (Dutch version)).

OTHER OUTCOMES:
Intensity of non-residential grandchild care | At baseline (T0), at 12 months (T1), at 24 months (T2)
  A self-reported questionnaire (only to be administered in the subsamples of grandparents) will be used to register specific information on the intensity of the non-residential grandchild care they provide in a typical week.
Socio-demographic characteristics | At baseline (T0), at 12 months (T1), at 24 months (T2)
  A self-reported questionnaire will be used to collect the necessary demographic information of the participants (i.e., date of birth, sex, marital status, and possible date of retirement), and (if applicable) of their grandchild(ren) (i.e., number of grandchildren, date of birth and the sex of each individual grandchild).

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided